CLINICAL TRIAL: NCT06828562
Title: GENomic Predictors in A Multi-Ethnic Population With Kidney Disease Study
Acronym: Genie
Status: Enrolling by invitation | Type: Observational
Sponsor: Western Sydney Local Health District (Other)
Responsible Party: Principal Investigator, Jennifer Li, Principal Investigator, Western Sydney Local Health District
Other Study IDs: GENIE Study
Record Dates: First submitted 2025-02-10; First posted 2025-02-14 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-02

CONDITIONS: Kidney Disease
Keywords: kidney
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Biospecimen Retention: Samples With DNA — Blood and or residual biopsy (archive) tissue Optional - urine and faecal samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Group 1 - Healthy participants (without established kidney disease): eGFR > 60ml/min/1.73m2, UACR < 3 mg/mmol (or UPCR < 10 mg/mmol)
  Has risk factors for kidney disease, including any of the following:
  Family history of kidney disease (CKD, dialysis or transplant) Any history of acute kidney injury or eGFR decline from baseline Established diabetes, hypertension, stroke, heart disease or heart failure Current or ex-smoker, overweight (BMI > 25) or obesity (BMI > 30)
- Group 2 - Participants with established chronic kidney disease (CKD): eGFR ≤ 60ml/min/1.73m2 (over minimum 3-month period), or UACR > 30mg/mmol (or PCR > 100mg/mmol). CKD can be from any cause/aetiology.
- Group 3 - Participants with kidney failure and are on dialysis: Patients established on peritoneal dialysis or haemodialysis for at least 3 months

SUMMARY:
To establish a prospective, longitudinal cohort of participants who can provide blood, tissue (including kidney histology), urine samples to establish a core biobank for kidney disease research. Results from this biobank will be matched to clinical outcomes to facilitate the discovery (and/or validation) of novel prognostic, predictive or diagnostic biomarkers important for kidney disease.

DETAILED DESCRIPTION:
Hypothesis:

Genetic ancestry influences the enrichment of certain polymorphisms, which may have important protective or adverse effects on important kidney related outcomes, including developing chronic kidney disease, progression to kidney failure, and/or poor long-term outcomes following kidney transplantation.

Aims:

To establish a prospective, longitudinal cohort of participants who can provide blood, tissue (including kidney histology), urine samples to establish a core biobank for kidney disease research. Results from this biobank will be matched to clinical outcomes to facilitate the discovery (and/or validation) of novel prognostic, predictive or diagnostic biomarkers important for kidney disease. Data from this cohort will be used to determine if genomic factors independently influence:

1. The susceptibility to developing acute kidney injury (AKI) and the severity of AKI.
2. The development of chronic kidney disease (CKD), and the complications of CKD
3. The progression to kidney failure (needing dialysis or transplant) and complications of kidney failure?
4. The risk of treatment failure (or resistance) to standard medical therapy for any of the above (1-4)?

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old at time of enrolment
* Able to provide consent
* Either have kidney disease at time of enrolment or not have kidney disease but has at least one risk factor for kidney disease (eg family history, hypertension, diabetes, smoking, stones, nephrotoxin use)
* Consent to longitudinal follow up at enrolment
* Consent to providing blood samples at enrolment

Exclusion Criteria:

* Unable or unwilling to provide consent
* life-expectancy less than 6-months
* received haematopoietic stem cell transplant in the past 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Australian participants - health and kidney disease (groups described earlier)
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2040-01-01 (Estimated); Study Completion 2050-01-01 (Estimated)

PRIMARY OUTCOMES:
Development of CKD | 20 years
  Group 1 develops eGFR ≤ 60ml/min/1.73m2 (or biopsy proven kidney disease) ≥ 3-months, or albuminuria or proteinuria (UACR > 3mg/mmol or UPCR > 10mg/mmol) ≥ 3-months
Progression of CKD | 20 years
  For group 2, defined by eGFR decline ≥ 30% from baseline for ≥ 3 months, or eGFR decline to below 15ml/min/1.73m2 if baseline eGFR > 30ml/min/1.73m2, or the need for renal replacement therapy
Removal from dialysis | 20 years
  For group 3 - either death (survival time on dialysis) if they do not receive a kidney transplant during the study, or if they receive a kidney transplant

SECONDARY OUTCOMES:
Death | 20 years
  death from any cause
Hospital Admissions | 20 years
  Hospital or emergency department visits for any reason
estimated glomerular filtration rate slope | 10 and 20 year time points
  change in eGFR over time
Cardiovascular event or major risk factors | 20 years
  (MACE): non-fatal stroke, non-fatal myocardial infarction, cardiovascular death. Major risk factors: diabetes mellitus, dyslipidaemia, obesity, hypertension
Major infectious events | 20 years
  bacterial, fungal or viral infection which necessitates hospital admission or medical attention
Malignancy | 20 years
  any cancer diagnosis following enrolment
acute kidney episodes | 20 years
  acute kidney episodes (defined by KDIGO criteria), registry code or clinician assignment for group 1 or 2
Dialysis dose | 10 years
  time on dialysis (hours/days) and dialysis prescription (if available)

CONTACTS AND LOCATIONS:
Locations (4):
- Australia (4):
  - Royal Prince Alfred Hospital, Sydney, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Westmead Institute for Medical Research, Westmead, New South Wales
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: No
Confidential information and data sharing requires additional ethics submission or individual participant consent